CLINICAL TRIAL: NCT04099602
Title: Investigation of the Effect of Massage on Bilirubin Level in Preterm Infants
Brief Title: The Effect of Massage on Bilirubin Level in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gönül Kılıç, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EgeU
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Massage; Neonatal Jaundice
Keywords: neonatal jaundice; baby massage; transcutaneous bilirubin level; premature infant
MeSH Terms: conditions — Jaundice, Neonatal; Premature Birth

STUDY DESIGN:
Intervention Model Description: In the study, the investigators were decided that at least 30 premature infants were included in each group considering that losses might occur during data collection. Block randomization method was used to control the selection bias that might arise during the determination of the study groups. In this method, the number and probability of groups are equal in each block. Infants in both groups were randomized to block stratified by sex and gestational week. In the block randomization, blocks are selected randomly and this process is continued until all the subjects to be included in the study are assigned to the groups and the number of subjects in the groups is equalized at the end of this procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Experimental): Twice a day after the birth of the baby was massaged by the researcher for 5 days. Bilirubin levels were measured twice daily by the transcutaneous bilirubin meter before the morning massage and 2 hours after the evening massage for 5 days. In the morning (between 07:00-09:00 am) and in the evening (between 19:00-21:00 pm) twice a day, 15-20 minutes baby massage was applied.
  Interventions: Other: Baby Massage
- Control group (No Intervention): The control group who were administered standard care and bilirubin levels were measured twice daily by the transcutaneous bilirubin meter for 5 days

INTERVENTIONS:
Other: Baby Massage — Received baby massage and bilirubin levels were measured twice daily by the transcutaneous bilirubin meter for 5 days
  Arms: Massage group

SUMMARY:
Jaundice (hyperbilirubinemia) which is one of the common causes of repeated hospitalizations in the neonatal period, is a physiological condition seen in 60% of term babies and 80% of premature babies in the first week of life . Premature babies are more susceptible tobilirubin neurotoxicity. Death and severe sequelae due to hyperbilirubinemia can be prevented by early diagnosis and treatment. Massage is one of the applications that can be used to reduce bilirubin levels in newborn infants. Baby massage facilitates bowel movements and bilirubin excretion by reducing enterohepatic circulation. This study was designed as a randomized controlled trial to investigate the effect of massage on bilirubin levels in premature infants.

DETAILED DESCRIPTION:
Neonatal jaundice is a physiological condition seen in 60% of infants and 80% of preterm infants in the first week of life. There is no clear data on the frequency of jaundice in newborns in our country. Jaundice is one of the common causes of 75% of hospitalizations in the first week after birth and the recurrence of hospitalizations in the neonatal period. Neonatal jaundice is a non-hazardous and transient condition that can usually resolve spontaneously without treatment. Although it is a transient condition, high bilirubin levels can cause kernicterus which causes severe neurological damage if not diagnosed and treated early .

The severity and complications of hyperbilirubinemia in premature infants are different from term infants. Premature infants are more susceptible to damage caused by serum bilirubin, even at low levels of brain cells. Hyperbilirubinemia in preterm infants is more prevalent, severe, and protracted than that in term infants because of the immaturity of their red blood cells, livers, and gastrointestinal tracts. There also is often a delay in enteral feeds, which may limit intestinal flow and bacterial colonization, resulting in further enhancement of the enterohepatic circulation of bilirubin. Preterm neonates are more susceptible to bilirubin neurotoxicity. Almost all preterm infants less than 35 weeks gestational age have elevated total serum/plasma bilirubin levels, which results in neonatal jaundice, the yellowish discoloration of the skin and conjunctiva caused by bilirubin deposition. The major complication of an elevated total serum (hyperbilirubinemia) is bilirubin-induced neurologic dysfunction (BIND), which occurs when circulating bilirubin crosses the blood-brain barrier and binds to brain tissue . Jaundice is an important problem in newborn infants and death and severe sequelae due to hyperbilirubinemia can be prevented by early diagnosis and treatment. Various treatment methods have been developed to reduce bilirubin levels. The most commonly used methods are; blood exchange, phototherapy and pharmacological agents. Therapeutic interventions prevent BIND and thus kernicterus by lowering the level of bilirubin in the blood. Phototherapy is a common treatment for both treatment and prevention of increased bilirubin levels. Phototherapy has been widely used in the treatment of hyperbilirubinemia of the newborn for more than fifty years. Phototherapy has various side effects, such as damage to the retina and genitalia, loss of body water, skin rashes, watery stools and Bronze Baby Syndrome.

Nowadays, studies on new treatment methods and different applications are being made which support the treatment of jaundice and shorten the length of hospital stay. Kangaroo care reduces the exposure of newborns to phototherapy, swimming, wiping and bathtub bathing have been reported to reduce bilirubin levels. Baby massage is one of the alternative and complementary therapies that can be used to reduce bilirubin levels.

While there are many studies investigating the effect of infant massage on bilirubin levels in term neonates with healthy and hyperbilirubinemia, a limited number of studies investigating the effect of massage on bilirubin levels in premature infants were found.

It is suggested that baby massage can be performed by trained nurses and mothers trained by nurses. Infant massage stimulates defecation by increasing bowel movements, thus decreasing enterohepatic circulation and increasing bilirubin excretion. Bilirubin excretion decreases the speed and severity of hyperbilirubinemia. In some studies investigating the effect of massage on bilirubin levels, transcutaneous bilirubin (TcB) levels or TSB levels were found to be significantly lower, also no significant difference was found in some studies.

In our country, the studies on the benefits of baby massage for infants are quite new. There are two studies investigating the effect of massage on bilirubin levels in newborn infants. However, in one of these studies, the effect of infant massage on bilirubin levels in newborns who received phototherapy was investigated, while the effect of abdominal massage on TcB bilirubin levels in newborns was investigated in the other study. TSB levels are the gold standard in the evaluation of bilirubin levels in newborn infants. However, the blood needs to be taken from the baby, and taking blood is a painful procedure, and it may not always possible to get enough blood. Measurement of bilirubin level from the skin surface is both noninvasive, painless and simple. In this study, the effect of infant massage on bilirubin level in premature infants not receiving phototherapy was evaluated by transcutaneous bilirubin measurement method. This study was designed as a randomized controlled trial to investigate the effect of massage on bilirubin levels in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* families being voluntary to participate in the study
* infants being born between 32 and 37 weeks plus 6 days of gestation
* infants having a birth weight of ≥1500 g
* infants having a fifth-minute Apgar score of more than seven
* infant's bilirubin level is not sufficient to require phototherapy
* the vital signs of the baby are within normal limits
* the absence of congenital major malformation of the infants
* the lack of patent ductus arteriosus requiring treatment
* no proven sepsis diagnosis

Exclusion Criteria:

* neonates with disease disrupting skin integrity (epidermolysis bullosa, ichthyosis, collodion baby)
* need for phototherapy
* infants with gastrointestinal obstruction and biliary atresia
* infants with congenital major deformations

Ages: 32 Weeks to 38 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Transcutaneous Bilirubin Levels | "through study completion, an average of 1 year"
  bilirubin level mg/dl

SECONDARY OUTCOMES:
frequency of defecation | "through study completion, an average of 1 year"
  daily number

OTHER OUTCOMES:
length of hospital stay | "through study completion, an average of 1 year"
  number of days in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Bal Yılmaz, Prof., Study Director — Ege University
Locations (1):
- Ege University Faculty of Nursing, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No